CLINICAL TRIAL: NCT03730532
Title: Comparing Cognitive-behavioural and Cognitive-analytic Guided Self-help for Anxiety; a Patient Preference Clinical Trial
Brief Title: Guided Self-help for Anxiety - a Patient Preference Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Emma Beattie-Edwards, Trainee Clinical Psychologist, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240751
Record Dates: First submitted 2018-10-16; First posted 2018-11-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Anxiety
Keywords: Guided self help; Cognitive Analytic Therapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patient Preference Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomised CBT (Experimental): Cognitive Behavioural Therapy Guided Self Help
  Interventions: Other: Cognitive Behavioural Therapy Guided Self Help
- Randomised CAT (Experimental): Cognitive Analytic Therapy Guided Self Help
  Interventions: Other: Cognitive Analytic Therapy Guided Self Help
- Preference CAT (Experimental): Cognitive Analytic Therapy Guided Self Help
  Interventions: Other: Cognitive Analytic Therapy Guided Self Help
- Preference CBT (Experimental): Cognitive Behavioural Therapy Guided Self Help
  Interventions: Other: Cognitive Behavioural Therapy Guided Self Help

INTERVENTIONS:
Other: Cognitive Behavioural Therapy Guided Self Help — 6-week manualised Cognitive Behavioural Therapy Guided Self Help
  Arms: Preference CBT; Randomised CBT
Other: Cognitive Analytic Therapy Guided Self Help — 6-week manualised Cognitive Analytic Therapy Guided Self Help
  Arms: Preference CAT; Randomised CAT

SUMMARY:
Supporting patients in exerting choice over their treatment is a central aspect of modern healthcare. In Improving Access to Psychological Therapies (IAPT) services, then patients treated at step 2 are only and always offered cognitive-behaviourally informed guided self-help (GSH), when they are deemed suitable for treatment at step 2 of IAPT services (termed CBT-GSH). Step 2 interventions are guided self-help (GSH) delivered by Psychological Wellbeing Practitioners (PWPs). Recently, a new type of GSH has been developed and found to be feasible and effective in IAPT services - this is called cognitive-analytic guided self-help (CAT-GSH). This research aims to test the efficacy of CAT-GSH by comparing outcomes over time achieved in both types of GSH and interviewing participants about their experience of the GSH. The methodology to support patient choice is a patient preference trial. In this method, then patients that meet inclusion criteria for the trial are offered and choose between either CAT-GSH and CBT-GSH. Those patients that are unconcerned with the type of treatment are randomised to either CAT-GSH or CBT-GSH. The primary outcome measure is the Beck Anxiety Inventory. No changes to the standard practice of the PWPs will occur during the trial, the trial will be situated in a standard IAPT service and be a therefore conducted in a routine practice setting.

ELIGIBILITY:
Inclusion Criteria:

* patients have self-referred or been referred by their GP or other health or social care professional for a step 2 intervention for treatment of a common mental health problem,
* patients meet criteria for an anxiety disorder on MINI screening interview assessment and also met caseness on the BAI (as defined by a score of >10 on the BAI at assessment).
* Patients want to engage in GSH to address the anxiety disorder
* patients are motivated to engage in treatment and can attend six sessions of face-to-face GSH.

Exclusion Criteria:

* engaging in any another IAPT step 2 interventions.
* Do not meet criteria for an anxiety disorder as defined by the MINI and the BAI score.
* Meet criteria for depression and a comorbid anxiety disorder, as identified by the BAI and MINI, where the depression is more severe and is the patient's main concern.
* Have a severe/chronic mental health problem and are already involved in psychiatric or secondary care mental health services.
* Have substance misuse issues that would interfere with engagement with the GSH.
* Have a diagnosed learning disability that precludes engagement in GSH.
* Have a diagnosis of social phobia or PTSD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | Measured at screening, at 6 weeks, 12 weeks and 24 weeks
  measuring change in anxiety at four time points

SECONDARY OUTCOMES:
Generalised Anxiety Disorder - 7 | Measured at screening, weekly for 6 weeks, then at 12 week and 24 week follow-up
  measuring change in anxiety across the intervention and follow-up
patient health questionnaire - 9 | Measured at screening, weekly for 6 weeks, then at 12 week and 24 week follow-up
  measuring change in depression across the intervention and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Steve Kellett, Study Director — University of Sheffield
Locations (1):
- Oldham Healthy Minds IAPT, Oldham, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kellett S, Bee C, Smithies J, Aadahl V, Simmonds-Buckley M, Power N, Dugen-Williams C, Fallon N, Delgadillo J. Cognitive-behavioural versus cognitive-analytic guided self-help for mild-to-moderate anxiety: a pragmatic, randomised patient preference trial. Br J Psychiatry. 2023 Sep;223(3):438-445. doi: 10.1192/bjp.2023.78. PMID 37395600